CLINICAL TRIAL: NCT07071649
Title: Evaluation of a Plasma Marker (p-Tau217) for the Biological Diagnosis of Alzheimer's Disease, and Comparison With CSF Markers
Acronym: ALZBIOSANG
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PI2024_843_0128
Record Dates: First submitted 2025-07-08; First posted 2025-07-17 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Alzheimer's Disease; Biomarkers; Non-invasive Diagnosis; Phosphorylated Protein p-tau217
Keywords: Alzheimer's Disease; Biomarkers; Non-invasive diagnosis; Phosphorylated protein p-tau217
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: blood withdrawal — blood withdrawal

SUMMARY:
The biological diagnosis of AD is actually performed by analysing Aβ1-40 and Aβ1-42 peptides, total tau and tau phosphorylated at Thr181 (p-Tau181) from cerebrospinal fluid (CSF) samples obtained by lumbar puncture (LP). Phospho-Tau 217 (p-Tau217) is a new biomarker that could be measured in plasma. The aim of this study is to compare the performances of plasma p-Tau217 with those of the reference CSF biomarkers in 150 patients recruited in the memory center of CHU Amiens (France). The study will be conducted during 18 months. The inclusion will be proposed to all patients for whom an indication of lumbar puncture / CSF is raised in a context of clinical suspicion of AD. During the daily hospitalization during which CSF will be collected for the "classical" biomarkers testing, a single tube of blood will be collected (anticoagulant EDTA, collected for p-Tau 217 analysis). The performances of CSF and plasma pTau 217 will be compared with the clinical diagnosis of AD (+, -, or indeterminate).

ELIGIBILITY:
Inclusion Criteria:

* All patients addressed to the memory center of CHU Amiens with a clinical suspicion of AD, for whom lumbar puncture / CSF biomarkers of AD determination is proposed.

Exclusion Criteria:

* Minor patients
* pregnant women
* patients under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-11-20 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
plasma p-Tau217 concentration | day 1
  Analysis of performances of plasma p-Tau217 for the diagnosis of AD by using the kit supplier references.

SECONDARY OUTCOMES:
concordance of plasma-pTau217 with CSF biomarkers | day 1
  Comparison of plasma-pTau217 with CSF biomarkers, realization of a concordance matrix.

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No